CLINICAL TRIAL: NCT06510842
Title: Lumbar Drainage of Intraventricular Hemorrhage The DRAIN IVH Randomized Controlled Trial
Brief Title: Lumbar Drainage of Intraventricular Hemorrhage
Acronym: DRAIN IVH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Silvia Schönenberger, MD, Prof. Dr. Silvia Schönenberger, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRAIN IVH; S-304/2024 (Other: Medizinische Ethikkomission Heidelberg)
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Intraventricular Hemorrhage; Lumbar Drainage; External Ventricular Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Additional insertion of a lumbar drainage.
  Interventions: Other: External drainage of intraventricular hemorrhage
- Control arm (Active Comparator): Standard of care consists of drainage of CSF via EVD with or without intraventricular thrombolysis.
  Interventions: Other: External drainage of intraventricular hemorrhage

INTERVENTIONS:
Other: External drainage of intraventricular hemorrhage — An EVD is required to be eligible for the DRAIN IVH study. Weaning from the EVD is at the discretion of the local investigators. Imaging is at discretion of local investigators. Use, timing and frequency of fibrinolysis via EVD is at local discretion, too.

SUMMARY:
Intracerebral hemorrhage (ICH) is a debilitating and fatal disease, especially when the hemorrhage is also entering the cerebral ventricles leading to acute hydrocephalus. In these cases, patients need a drainage through external ventricular drains (EVD). In the longer term, patients often need a permanent ventriculoperitoneal (VP) shunt to avoid hydrocephalus. Here we hypothesize that the early insertion of a lumbar drainage in addition to the EVD could lead to better functional outcome and avoidance of VP shunting by drainage of the blood which promotes inflammatory and adverse effects in the subarachnoid space. For that we propose a multi-center randomized clinical trial to investigate the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* ICH with IVH (with hemorrhage in the 3rd and/or 4rth ventricle) with the need for EVD placement due to acute hydrocephalus
* Age ≥ 18 y
* Lumbar drain can be inserted within 72 h after symptom onset or patient last seen well

Exclusion Criteria:

* Premorbid mRS score > 2
* Pregnancy
* Life expectancy <6 months
* Patient/family/caregiver unwilling or unlikely to opt for at least two weeks of aggressive therapy prior to consideration of transition to comfort measures/discontinuation of life support measures.
* Treating physicians deeming the prognosis as so grave that an aggressive therapy is not warranted.
* Other clear contraindication for treatment with a lumbar drain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Rate of mRS | 180 days (+/- 14 days)
  The mRS is frequently employed to assess functional outcome of stroke therapy - its ease of use, simplicity of interpretation for clinicians and families, and agreement with other stroke scales are appealing features. The use of fixed dichotomous analysis of ordered categorical outcomes after stroke (mRS 0-3 favorable vs. 4-6 non-favorable outcome) has proved to be valid and reliable for defining outcome in stroke patients in many previous studies.

SECONDARY OUTCOMES:
Amount of CSF drained by external ventricular drain | up to 14 days (duration of hospital stay)
  in ml
Amount of CSF drained by lumbar drain | up to 14 days (duration of hospital stay)
  in ml
Need for VP shunt | up to 14 days (duration of hospital stay)
  operative implantation of VP shunt
Need for VP shunt | at 180 days
  operative implantation of VP shunt
Clearance of intraventricular blood (via neuroimaging with CT or MRI) | up to 14 days (duration of hospital stay)
  Opening of third ventricle (y/n)
Clearance of intraventricular blood (via neuroimaging with CT or MRI) | up to 14 days (duration of hospital stay)
  Opening of fourth ventricle (y/n)
Bacterial Ventriculitis/Meningitis leading to antibiotic treatment | up to 14 days (duration of hospital stay)
  (y/n)
Mortality | up to 14 days (duration of hospital stay) and 6 month
  cerebral cause of death (y/n)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Schönenberger, MD, Principal Investigator — Heidelberg University Hospital, Department of Neurology
Locations (12):
- Germany (12):
  - Department of Neurology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - LMU München, München, Bavaria
  - Augsburg University Hospital, Augsburg
  - Charite Universitätsmedizin Berlin, Berlin
  - Düsseldorf Universitiy Hospital, Düsseldorf
  - Frankfurt University Hospital, Frankfurt
  - Goettingen University Hospital, Göttingen
  - Augsburg University Hospital Department of Neurosurgery, Heidelberg
  - Heidelberg University Hospital Department of Neurosurgery, Heidelberg
  - Mainz University Hospital, Mainz
  - Mannheim University Hospital, Mannheim
  - Osnabrück Clinic, Osnabrück

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Staykov D, Kuramatsu JB, Bardutzky J, Volbers B, Gerner ST, Kloska SP, Doerfler A, Schwab S, Huttner HB. Efficacy and safety of combined intraventricular fibrinolysis with lumbar drainage for prevention of permanent shunt dependency after intracerebral hemorrhage with severe ventricular involvement: A randomized trial and individual patient data meta-analysis. Ann Neurol. 2017 Jan;81(1):93-103. doi: 10.1002/ana.24834. PMID 27888608
- [Background] Staykov D, Huttner HB, Struffert T, Ganslandt O, Doerfler A, Schwab S, Bardutzky J. Intraventricular fibrinolysis and lumbar drainage for ventricular hemorrhage. Stroke. 2009 Oct;40(10):3275-80. doi: 10.1161/STROKEAHA.109.551945. Epub 2009 Aug 13. PMID 19679848
- [Background] Kuramatsu JB, Gerner ST, Ziai W, Bardutzky J, Sembill JA, Sprugel MI, Mrochen A, Kolbl K, Ram M, Avadhani R, Falcone GJ, Selim MH, Lioutas VA, Endres M, Zweynert S, Vajkoczy P, Ringleb PA, Purrucker JC, Volkmann J, Neugebauer H, Erbguth F, Schellinger PD, Knappe UJ, Fink GR, Dohmen C, Minnerup J, Reichmann H, Schneider H, Rother J, Reimann G, Schwarz M, Bazner H, Classen J, Michalski D, Witte OW, Gunther A, Hamann GF, Lucking H, Dorfler A, Ishfaq MF, Chang JJ, Testai FD, Woo D, Alexandrov AV, Staykov D, Goyal N, Tsivgoulis G, Sheth KN, Awad IA, Schwab S, Hanley DF, Huttner HB; Collaborators. Association of Intraventricular Fibrinolysis With Clinical Outcomes in Intracerebral Hemorrhage: An Individual Participant Data Meta-Analysis. Stroke. 2022 Sep;53(9):2876-2886. doi: 10.1161/STROKEAHA.121.038455. Epub 2022 May 6. PMID 35521958